CLINICAL TRIAL: NCT05968274
Title: The Effect of Rebox Current in Pain Management
Acronym: REBOX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rebox Therapy s.r.o. (Industry)
Collaborators: F.D. Roosevelt University Hospital in Banská Bystrica, Slovakia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14/2023
Record Dates: First submitted 2023-07-15; First posted 2023-08-01 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Electric Stimulation Therapy
Keywords: Rebox therapy; electrotherapy; pain treatment; Rebox currents
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm "A" (Other): 1. First stimulation period: real stimulation, total 8 sessions, session frequency: weekdays every other day (i.e. duration 2.5 weeks)
  2. Washout period: no stimulation, duration: 1 week
  3. Second stimulation period: sham stimulation, total 8 sessions, session frequency: weekdays every other day (i.e. duration 2.5 weeks)
  Interventions: Device: Rebox-Physio 4 (real stimulation); Device: Rebox-Physio 4 (sham stimulation)
- Arm "B" (Other): 1. First stimulation period: sham stimulation, total 8 sessions, weekdays every other day (i.e. 2.5 weeks)
  2. Washout period: no stimulation, 1 week
  3. Second stimulation period: real stimulation, total 8 sessions, weekdays every other day (i.e. 2.5 weeks)
  Interventions: Device: Rebox-Physio 4 (real stimulation); Device: Rebox-Physio 4 (sham stimulation)

INTERVENTIONS:
Device: Rebox-Physio 4 (real stimulation) — Rebox-Physio 4 is a CE-certified medical device class IIa. The device is a voltage-controlled generator of specific DC electric pulses with voltage amplitude 0-21 V, current intensity up to 200 uA, rectangular pulse shape, pulse frequency 3000 Hz and pulse duration 0.25 ms. Rebox currents are applied locally at the site of pain non-invasively transcutaneously with a touch of a flexible pin active treatment electrode (cathode) while the patient holds a cylindrical electrode (anode) to close electric circuit. Stimulation time in one point is 3-5 seconds until the current intensity reaches stable target values of 140-160 uA. During one session, total 20-50 points are systematically treated at a mutual distance of approx. 2 cm over the target region.
Device: Rebox-Physio 4 (sham stimulation) — In the sham stimulation, the comparator will be a visually identical sham version of the real Rebox-Physio 4.The sham device has a resistor installed at the output generating current of negligible intensity (maximum 1 uA) assuming no relevant physiological effect. The application procedure will be identical to the real device. When applied to the patient, the sham device displays "false" voltage and current intensity values and responds to the operator´s actions in real time mimicking the real stimulation. The operator is therefore blinded.

SUMMARY:
This post-marketing monocentric double-blind sham controlled crossover study will assess the efficacy of Rebox electrotherapy in the treatment of pain. Totally 72 patients will be treated with both real and sham Rebox device in a crossover design with a 1:1 ratio over a 6-week period. The degree of pain intensity reduction after the real Rebox stimulation will be evaluated in comparison with the sham stimulation. Moreover, differences in multidimensional aspects of pain will be compared between the real and sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with pain based on the following diagnoses:

  * Myofascial musculoskeletal pain
  * Vertebrogenic algic syndrome in the cervical, thoracic and lumbosacral regions
  * Sacroileitis with sacroiliac joint block
  * Cervicocranialgia
  * Frozen shoulder syndrome
  * Arthrosis
  * Epicondylitis
  * Pain in tendons, ligaments and other enthesopathies
  * Postoperative pain
  * Post-traumatic pain
  * Postherpetic neuralgia
* Duration of pain (de novo or exacerbation of chronic pain) prior to study inclusion ranges from 2 weeks to 3 months
* The average pain intensity in a given period of 2 weeks to 3 months prior to study inclusion must be NRS (Numerical Rating Scale) >3
* The patient may be concurrently treated with analgesics and may be undergoing manual physiotherapy (rehabilitation)

Exclusion Criteria:

* Age <18 years
* Local contraindications:

  * Impaired skin integrity at the site of application (open wound, skin ulcer, burns), Note: the area around the postoperative scar is not an exclusion criterion
  * Acute inflammation of the skin or subcutaneous tissue at the application site
  * Deep vein thrombosis (diagnosed or suspected)
* General contraindications:

  * Implanted electrical device (pacemaker, implantable cardioverter-defibrillator, deep brain stimulator, cochlear implant, etc.)
  * Pregnancy
  * Epilepsy
  * Malignant cancer (diagnosed or suspected)
  * Acute potentially life-threatening conditions
* Concomitant other physical therapy (electrotherapy, magnetotherapy, laser therapy, ultrasound therapy, mechanotherapy, etc.)
* The Rebox device was administered to the subject for any indication in the last 12 months prior to the study inclusion date
* A recent change in analgesic medication (i.e., new agent or change in agent dose less than 1 week prior to the first stimulation session) or a planned change in analgesic medication during the course of the study (change in agent, change in dose), Note: modification of analgesic medication during the study is possible but must be recorded
* Ongoing acute infection, surgery or trauma during the study
* Concurrent subject participation in another clinical study
* Subject is unable to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity | 1. at baseline (day of randomization); 2. after 8th session (at the end of week 2.5 from randomization); 3. before 9th session (at the end of week 3.5 from randomization); 4. after 16th session (at the end of week 6 from randomization)
  The degree of change in pain intensity after the real vs. sham stimulation will be evaluated between 4 specified time points. The Numerical Rating Scale (NRS) will be used to assess pain intensity. Pain scores will be assessed by completing the Brief Pain Inventory (BPI).

SECONDARY OUTCOMES:
Immediate analgesic effect | At each stimulation session, total 16 times (at 8 weekdays every other day from randomization up to week 2.5 + at 8 weekdays every other day from week 3.5 up to week 6)
  The trend of the intra-individual effect of the real vs. sham stimulation on immediate pain relief will be assessed. The Numerical Rating Scale (NRS) will be used to assess pain intensity.
Change in multidimensional aspects of pain | 1. at baseline (day of randomization); 2. after 8th session (at the end of week 2.5 from randomization); 3. before 9th session (at the end of week 3.5 from randomization); 4. after 16th session (at the end of week 6 from randomization)
  The degree of change in multidimensional aspects of pain after the real vs. sham stimulation will be evaluated between 4 specified time points. Items related to multidimensional aspects of pain will be included in the BPI questionnaire (items 9 a-g).
  The degree to which pain affects the following aspects will be assessed (in tens of %).
  1. Activity in general
  2. Mood
  3. Ability to walk
  4. Normal work (including work outside the home and housework)
  5. Relationships with other people
  6. Sleep
  7. Enjoyment of life
Tolerability outcome | At each stimulation session, total 16 times (at 8 weekdays every other day from randomization up to week 2.5 + at 8 weekdays every other day from week 3.5 up to week 6)
  The percentage of patients who complete the entire study will be determined. The application will be considered well tolerated by the patient if a minimum of 14 out of 16 sessions are completed. Overall, the application will be considered well tolerated if tolerated application is achieved in ≥ 90% of patients without the need for early discontinuation due to intolerance. Any technical complications/adverse effects during application will be recorded in the application protocol and will be analyzed by the study monitor at a minimum interval of once per month .

CONTACTS AND LOCATIONS:
Overall Officials: Igor Martuliak, MD, PhD, Principal Investigator — F.D. Roosevelt University Hospital in Banská Bystrica, Slovakia
Locations (1):
- F.D. Roosevelt University Hospital, Banská Bystrica, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Low J, Reed A. Electrotherapy Explained, Principles and Practice, 3rd Edition. Butterworth-Heinemann. 2000; 121-122.
- [Background] Johannsen F, Gam A, Hauschild B, Mathiesen B, Jensen L. Rebox: an adjunct in physical medicine? Arch Phys Med Rehabil. 1993 Apr;74(4):438-40. PMID 8466428
- [Background] Trudel D, Duley J, Zastrow I, Kerr EW, Davidson R, MacDermid JC. Rehabilitation for patients with lateral epicondylitis: a systematic review. J Hand Ther. 2004 Apr-Jun;17(2):243-66. doi: 10.1197/j.jht.2004.02.011. PMID 15162109
- [Background] Daut RL, Cleeland CS, Flanery RC. Development of the Wisconsin Brief Pain Questionnaire to assess pain in cancer and other diseases. Pain. 1983 Oct;17(2):197-210. doi: 10.1016/0304-3959(83)90143-4. PMID 6646795
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245